CLINICAL TRIAL: NCT04736329
Title: Telmisartan Versus Enalapril in Heart Failure With Reduced Ejection Fraction Patients With Moderately Impaired Kidney Functions. "TRIUMF Trial"
Brief Title: Telmisartan Versus Enalapril in Heart Failure With Reduced Ejection Fraction Patients With Moderately Impaired Kidney Functions
Acronym: TRIUMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Lecturer of Cardiology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-352-2020
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telmisartan (Active Comparator): Telmisartan (20 up to 80mg) for RAAS inhibition, as part of their heart failure therapy.
  Interventions: Drug: Telmisartan
- Enalapril (No Intervention): Enalapril (2.5 up to 20mg ) for RAAS inhibition, as part of their heart failure therapy.

INTERVENTIONS:
Drug: Telmisartan — Telmisartan (20 up to 80mg) for RAAS inhibition, as part of heart failure therapy.
  Arms: Telmisartan

SUMMARY:
Heart Failure (HF) poses a major health burden in various populations, with devastating annual rates of morbidity and mortality. It is estimated that 1%-to-2% of the general population suffer from the heart failure syndrome.

HF with reduced ejection fraction (HFrEF) is the most studied among different strata of ejection fractions (compared to HFpEF and HFmrEF), and thus therapies with evidence based survival benefit are well identified.

The syndrome of heart failure and the subsequent reduced cardiac output triggers activation of neurohormonal compensatory responses aiming to augment cardiac output and tissue perfusion, like upregulation of sympathetic nervous system and over-activation of the Renin Angiotensin Aldosterone System. Nevertheless, overshooting of such compensatory mechanisms have deleterious effects on heart failure in terms of aggravation of symptoms and reduction of survival.

Angiotensin II acts primarily on type I receptors inducing the following:

* intense arteriolar vasoconstriction
* stimulates sodium reabsorption in the proximal convoluted tubules
* stimulates adrenal medulla to secrete catecholamines
* stimulates sympathetic nervous system, through facilitation of ganglionic stimulation
* modestly inhibits vagus (parasympathetic system)
* stimulates secretion of vasopressin/anti-diuretic hormone
* stimulates adrenal cortex to secrete aldosterone, which promotes sodium and water reabsorption and promotes potassium secretion at the distal convoluted tubules in addition to induction of myocardial remodeling and fibrosis
* constricts the glomerular efferent arteriole which increase filtration pressure and promotes proteinuria and nephron injury/loss.

While, angiotensin type II receptors activation have beneficial effects like vasodilatation and promoting endothelial function.

Accordingly, angiotensin converting enzyme inhibitors (ACEi), angiotensin-II receptor type I blockers (ARBs) or Angiotensin receptor blocker- neprilisin inhibitor (ARNI) are considered a cornerstone in HFrEF therapy for both: symptoms relief and improvement of survival. Yet, hypotension, hyperkalemia or worsening of renal function are potential side effects that occasionally may lead to ACEi/ARBs/ARNI intolerance and subsequent discontinuation with loss of their cardioprotective effects.

On the other hand, cardiorenal syndrome is a recently introduced medical category due to the frequent association of cardiac and renal dysfunction in clinical practice. CardioRenal Syndrome CRS type I; acute cardiac dysfunction leading to renal dysfunction, is reported in 25%-to-33% of acute heart failure patients, and this prevalence jumps to 70% in cases of cardiogenic shock. CRS type II; chronic cardiac dysfunction leading to renal dysfunction, was found in 45% of chronic heart failure patients.

Despite the definite renoprotective and antiproteinuric effects of RAAS blockade in patients with chronic renal impairment, in cases when the glomerular filtration is critically dependent on angiotensin II-mediated efferent vasoconstriction such as in patients with heart failure and severe depletion of circulating volume-, ACEi/ARBs can lead to profound reduction of the glomerular filtration rate (GFR). The concerns about the safety of RAAS blockade in the presence of renal impairment has led to profound underutilization of these drugs in CHF patients with renal impairment.

The very prevalent co-existence of heart failure and renal impairment prominently impairs patients' outcomes both by direct disease effects and indirectly due to the occasional but frequent enforced discontinuation of therapies with proven survival benefit.[6]

Telmisartan is an ARB with peculiar pharmacodynamic properties. Unlike most of the ACEi/ARBs family, Telmisartan primarily depends on hepatic excretion and only a minority depends on renal excretion. Telmisartan has been proved in human and animal studies to be an effective agonist of the peroxisome proliferator-activated receptor gamma (PPAR ɣ) which potentiates its renoprotective effects being acting by dual mechanism.

So, it can be hypothesized that Telmisartan might be better tolerated than standard ACEi/ARBs in HF patients with moderate renal impairment, guranteeing less frequent interruptions and more consistent cardioprotective and renoprotective effects. However, there is no wealth of data to support or deny this theory.

DETAILED DESCRIPTION:
Population of study & disease condition Chronic heart Failure patients with reduced ejection fraction, (LVEF <40%) associated with moderate impairment of renal functions, (eGFR by Cockroft-Gold equation 60-40 ml/min/m2).

Patients will be randomized to receive either Enalapril (2.5 up to 20mg ) or Telmisartan (20 up to 80mg) for RAAS inhibition, as part of their heart failure therapy.

Objectives:

- Compare efficacy, safety and tolerability of Telmisartan versus Enalapril in HFrEF patients with impaired renal function.

• Methodology in details: HFrEF patients with moderate renal impairment as defined per protocol and after accepting participation to the study, will be randomly allocated into 2 equal groups using closed envelopes randomization system based on web-based randomization tables. Group 1 will receive Enalapril (between 2.5 to 20mg daily) as tolerated. Group 2 will receive Telmisartan (between 10 to 80mg daily) as tolerated. Both groups will receive other guidelines directed medical therapy for HFrEF. Patients will be monitored for :-

* Improvement of NYHA class.
* Six-minutes walk test at baseline at 2, 6 and 12 months.
* Trends of changes in NT-BNP values from baseline and every 6 months.
* Changes in left ventricular dimensions and ejection fraction assessed by echocardiography at baseline, at 6 and 12 months.
* Rates of worsening kidney functions assessed by changes in serum creatinine and in eGFR from baseline.
* Rates of improvement in albuminuria and serum albumin assessed by urinary Albumin/Creatinine ratio and serum albumin levels respectively, at baseline at 2, 6 and 12 months.
* Rates of discontinuation of / intolerance to the used agent for RAAS inhibition (enalapril/telmisartan)
* Rates of rehospitalization for decompensated heart failure.
* Rates of rehospitalization for any reason.
* Cardiac death.
* All-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients with signs and/or symptoms of heart failure NYHA II, III or IV, with echocardiographic diagnosis of HFrEF..
* Moderate impairment of renal functions, assessed by measuring serum creatinine levels then estimating the glomerular filtration rate (eGFR) by Cockroft-Gold equation to be (60-40 ml/min/m2).

Exclusion Criteria:

* Refusal to participate in the study.
* Known allergy to enalapril/telmisartan components.
* Pregnant and lactating ladies.
* Severe renal impairment defined as eGFR<30ml/min/m2 at time of enrollment to the study.
* Known cases of bilateral severe renal artery stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
change in Six-minutes walk test | After 6 months
  Six-minutes walk distance between the 2 groups
Rate of occurrence of worsening renal function | through 2 months
  Worsening kidney functions assessed by change of eGFR from baseline.
Rates of discontinuation of- or intolerance to the used agent for RAAS inhibition (enalapril/telmisartan) | Through 6 months
  Rate of discontinuing Telmisartan or Enalapril in the corresponding group driven by side effects.

SECONDARY OUTCOMES:
Degree of improvement in albuminuria and serum albumin | After 6 months
  Assessment of urinary Albumin/Creatinine ratio and serum albumin levels
Rates of rehospitalization for decompensated heart failure. | Through 6 months
  Rates of rehospitalization for decompensated heart failure.
All-cause death. | Through 6 months
  Number of deaths occurring due to any cause in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy hospital, faculty of medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Samir A, Aboel-Naga S, Shehata A, Abdelhamid M. Telmisartan versus EnalapRil In heart failure with redUced ejection fraction patients with Moderately impaired kidney Functions; randomized controlled trial: "TRIUMF trial". Egypt Heart J. 2023 Aug 8;75(1):68. doi: 10.1186/s43044-023-00398-7. PMID 37552407